CLINICAL TRIAL: NCT00304239
Title: A Multicenter, Double Blind, Vehicle-controlled, Randomized Study of Photodynamic Therapy (PDT) With Metvix 160 mg/g Cream and Aktilite CL128 LED Light in Patients With Multiple Actinic Keratosis on the Face and/or Scalp
Brief Title: Metvix PDT Versus Vehicle PDT With Aktilite CL128 Lamp in Patients With Actinic Keratosis on the Face and Scalp
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PC T405/05; 2005-005015-13 (EudraCT Number)
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2022-08

CONDITIONS: Actinic Keratosis
Keywords: Methyl aminolevulinate; Photodynamic therapy; Aktilite CL128 LED light source; Multiple Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metvix-PDT (Experimental): Participants received Metvix-PDT (methyl aminolevulinate hydrochloride-Photodynamic therapy) 160 milligrams per gram (mg/g) cream on face and/or scalp for 3 hours on Day 0 and Day 7.
  Interventions: Combination Product: Metvix-PDT
- Vehicle-PDT (Placebo Comparator): Participants received Vehicle cream (Vehicle-PDT) on face and/or scalp for 3 hours on Day 0 and Day 7.
  Interventions: Combination Product: Vehicle-PDT

INTERVENTIONS:
Combination Product: Metvix-PDT — Metvix 160 mg/g Cream was applied for 3 hours with occlusive dressing, and illumination with non-coherent red light using the Aktilite CL128 lamp, with a total light dose 37 Joule/square centimeter (J/cm²). All eligible lesions on the participant were treated twice with an interval of 1 week between treatments.
  Arms: Metvix-PDT
Combination Product: Vehicle-PDT — Vehicle Cream was applied for 3 hours with occlusive dressing, and illumination with non-coherent red light using the Aktilite CL128 lamp, with a total light dose 37 J/cm². All eligible lesions on the participant were treated twice with an interval of 1 week between treatments.
  Arms: Vehicle-PDT

SUMMARY:
The purpose of this study was to compare the efficacy of Photodynamic Therapy (PDT) with methyl aminolevulinate (MAL) cream to PDT with vehicle cream, using the Light-emitting diode (LED) light source Aktilite CL128, in treatment of participants with multiple actinic keratosis (sun-damaged skin) on the face and/or scalp.

DETAILED DESCRIPTION:
Actinic keratoses are pre-malignant skin lesions, which may develop to squamous cell carcinomas (SCC). They are usually small, thin, erythematous, de-squamating lesions on light exposed atrophic skin and the lesions are often multiple.

Photodynamic therapy (PDT) is the selective destruction of abnormal cells through light activation of a photosensitiser in the presence of oxygen. These cells accumulate more photosensitiser than normal cells. The photosensitiser generates reactive oxygen species upon illumination.

For skin diseases, such as actinic keratosis (AK), there has been an increasing interest in using topically applied precursors of the photoactive porphyrins (PAP). The most commonly used precursors have been 5-aminolevulinic acid (ALA) and its derivatives. The present test drug contains methyl aminolevulinate, which penetrates the lesions well and shows high lesion selectivity.

Different light sources (i.e. CureLight, Aktilite CL16 and Aktilite CL128) had been used for the activation of PAP, which absorbs light in the range of 400-700 nanometer (nm). The present study used the Aktilite CL 128 lamp. Aktilite 128 was based on LED technology and emits a narrow red light spectrum with an average wavelength of 630 (+/-5) nm. This study was similar to two other studies performed, on which the U.S. approval of Metvixia cream was based except for the light source used. This study was one of two studies performed to document the safety and efficacy of the Aktilite CL 128 lamp when used in combination with Metvixia cream.

Previous studies have shown that the risks attributed to Metvixia PDT are few and related mainly to transient pain and local erythema during and shortly after treatment. These reactions are part of the expected local phototoxicity reaction. PDT offers an advantage to other treatment modalities for actinic keratosis, being a non-invasive treatment available on an outpatient basis. Several separate lesions can be treated simultaneously and the same lesion(s) can be treated repeatedly with success. There are no known systemic toxicity or interaction with other medication. The treatment is also lesion selective, leaving the surrounding tissue intact and functional, also allowing excellent cosmetic results after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of 4-10 previously untreated, not pigmented, non-hyperkeratotic AK lesions of 3 mm or more diameter of Grade 1 and/or 2 of the face and/or scalp where other therapies are unacceptable or considered medically less appropriate.
* Males or females above 18 years of age.
* Written informed consent.

Exclusion Criteria:

* Participants with porphyria.
* Participants immunosuppressed for idiopathic, disease specific or therapeutic reasons.
* Known allergy to MAL, a similar PDT compound or excipients of the cream.
* Participants with history of hypersensitivity to nut products or other known protein antigens.
* Participation in other clinical studies either currently or within the last 30 days.
* Participants receiving local treatment (including cryotherapy and curretage) in face / scalp area within the last 30 days.
* Participants receiving topical treatment (including imiquimod, 5-FU and diclofenac) in face / scalp area within the last 3 months.
* Pregnant or breast-feeding: All women of child-bearing potential must use adequate contraception (oral contraceptives, intrauterine device, contraceptive skin patch, etc) during the treatment period and one month thereafter. In addition, they must have a negative pregnancy test prior to treatment.
* Any conditions that may be associated with a risk of poor protocol compliance.
* Participants currently receiving regular ultraviolet radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2006-03-13 (Actual); Primary Completion 2007-01-23 (Actual); Study Completion 2007-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf M Szeimies, Professor, Principal Investigator — Klinik und Poliklinik für Dermatologie, Klinikum der Universität Regensburg
Locations (11):
- United States (4):
  - Ashish C. Bhatia, Naperville, Illinois
  - Joseph Fowler, Louisville, Kentucky
  - Robert T. Matheson, Portland, Oregon
  - Steven A. Davis, San Antonio, Texas
- Germany (7):
  - Hautklinik Heinrich Heine Universität, Düsseldorf
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt am Main, Frankfurt
  - Praxis Dr. Winfried Klövekorn, Gilching
  - Klinik für Dermatologie und Venerologie Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Klinikum der Universität München, Klinikum und Poliklinik für Dermatologie und Allergologie, München
  - Klinik und Poliklinik für Dermatologie, Klinikum der Universität Regensburg, Regensburg
  - Praxis Dr. Klemm, Tutzing

REFERENCES:
- [Background] Pariser DM, Lowe NJ, Stewart DM, Jarratt MT, Lucky AW, Pariser RJ, Yamauchi PS. Photodynamic therapy with topical methyl aminolevulinate for actinic keratosis: results of a prospective randomized multicenter trial. J Am Acad Dermatol. 2003 Feb;48(2):227-32. doi: 10.1067/mjd.2003.49. PMID 12582393
- [Background] Freeman M, Vinciullo C, Francis D, Spelman L, Nguyen R, Fergin P, Thai KE, Murrell D, Weightman W, Anderson C, Reid C, Watson A, Foley P. A comparison of photodynamic therapy using topical methyl aminolevulinate (Metvix) with single cycle cryotherapy in patients with actinic keratosis: a prospective, randomized study. J Dermatolog Treat. 2003 Jun;14(2):99-106. doi: 10.1080/09546630310012118. PMID 12775317

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 12 centers in Germany and the United States from 13 March 2006 to 23 January 2007.
Pre-assignment Details: A total of 131 participants were enrolled and received treatment in this study.
Period: Overall Study
Arm/Group | Metvix-PDT | Vehicle-PDT
Started | 73 | 58
Completed | 56 | 58
Not Completed | 17 | 0
Not completed — Protocol Deviations/Violations | 15 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: The safety population consisted of all participants for whom any kind of treatment was initiated.
Groups:
- Metvix-PDT: Participants received Metvix-PDT 160 mg/g cream on face and/or scalp for 3 hours on Day 0 and Day 7.
- Vehicle-PDT: Participants received Vehicle-PDT on face and/or scalp for 3 hours on Day 0 and Day 7.
- Total: Total of all reporting groups
Arm/Group | Metvix-PDT | Vehicle-PDT | Total
Number analyzed (Participants) | 73 | 58 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (8.4) | 67.0 (10.4) | 68.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 60 | 45 | 105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 73 | 58 | 131

OUTCOME MEASURES:

1. Primary Outcome: Participant Complete Response Rate (CRR)
Description: Participant complete response rate was defined as the percentage of participants with complete response. Complete response was defined as the complete disappearance of the lesion determined by clinical assessment (visual inspection and palpation) by an investigator.
Time Frame: At Week 13
Population: Intention-to-treat (ITT) population consisted of all participants that were randomized and for whom any aspect of treatment with either Metvix-PDT or Vehicle-PDT was initiated.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Metvix-PDT | Vehicle-PDT
Number analyzed (Participants) | 57 | 58
Percentage of participants | 68.4 [54.8 to 80.1] | 6.9 [1.9 to 16.7]

2. Secondary Outcome: Lesion Complete Response Rate
Description: Lesion complete response rate was defined as the percentage of pre-existing and treated lesions at baseline that were assessed as clear (complete disappearance of the lesion, visually and by palpation) after treatment. Percentage of lesions reported by location.
Time Frame: At Week 13
Population: as for outcome 1
Measure: Number; unit: Percentage of lesions
Units Other Than Participants: Lesion number
Arm/Group | Metvix-PDT | Vehicle-PDT
Number analyzed (Participants) | 57 | 58
Number analyzed (Lesion number) | 418 | 414
Percentage of lesions
  Face | 89 | 28
  Scalp | 81 | 30

3. Secondary Outcome: Number of Participants With at Least One Treatment Site Adverse Events
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily had a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. Number of participants with at least one treatment site adverse events were reported.
Time Frame: From start of study drug administration up to Week 13
Population: The safety population consisted of all participants for whom any kind of treatment was initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | Metvix-PDT | Vehicle-PDT
Number analyzed (Participants) | 73 | 58
Participants | 61 | 27

ADVERSE EVENTS:
Time Frame: From study drug administration up to Week 13
Description: The safety population consisted of all participants for whom any kind of treatment was initiated.
Groups:
- Vehicle-PDT: Participant received Vehicle-PDT 160 mg/g cream on face and/or scalp for 3 hours on Day 0 and Day 7.
Arm/Group | Metvix-PDT | Vehicle-PDT
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/58
Serious Adverse Events (participants affected / at risk) | 6/73 | 3/58
Other Adverse Events (participants affected / at risk) | 62/73 | 34/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metvix-PDT (N=73) | Vehicle-PDT (N=58)
Cerebral Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hospitalization for coronary cateterization (Investigations) | 1 (1) | 0 (0)
Basal cell carcinoma nose surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgery of squamous cell carcinoma right cheek (Surgical and medical procedures) | 1 (1) | 0 (0)
Re-surgery of squamous cell carcinoma right cheek (Surgical and medical procedures) | 1 (1) | 0 (0)
Lentigo maligna surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Planned three-step surgery of preexisting squamous cell carcinoma (Surgical and medical procedures) | 1 (1) | 0 (0)
Basal cell carcinoma left cheek surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Re-surgery and wound suture basal cell carcinoma left cheek (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee prothesis right due to arthrosis participants affected / exposed (Surgical and medical procedures) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Retrograde amnesia and anterograde amnesia due to cerebral concussion (Nervous system disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metvix-PDT (N=73) | Vehicle-PDT (N=58)
Pain of skin (Skin and subcutaneous tissue disorders) | 40 (40) | 12 (12)
Erythema (Skin and subcutaneous tissue disorders) | 38 (38) | 3 (3)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 26 (26) | 12 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (15) | 2 (2)
Skin discomfort (Skin and subcutaneous tissue disorders) | 10 (10) | 3 (3)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 11 (11) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 11 (11) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of participants analysed or technical problems leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes